CLINICAL TRIAL: NCT01914965
Title: A Randomized, Double-blind, Placebo-controlled Prospective Crossover Trial Investigating the Efficacy and Safety of the Treatment With Bupropion in Patients With Apathy in Huntington's Disease
Brief Title: Apathy Cure Through Bupropion in Huntington's Disease
Acronym: Action-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Ulm (Other); Ruhr University of Bochum (Other); University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Josef Priller, Prof. Dr. med. Josef Priller, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HDSY001; 2009-013698-16 (EudraCT Number)
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Apathy; Huntington's Disease
Keywords: Huntington's disease; Apathy; Bupropion
MeSH Terms: conditions — Lethargy; Huntington Disease | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Active Comparator): First treatment group: 150 mg bupropion or placebo once daily for 2 weeks, followed by 300 mg bupropion or placebo once daily for subsequent 8 weeks (until week 10; visit 4) First tapering and washout: 150 mg bupropion or placebo once daily for 7 days followed by a washout phase of 1 week on placebo
  Interventions: Drug: Bupropion; Drug: Placebo
- Placebo (Placebo Comparator): Second treatment group (crossover): placebo or 150 mg bupropion once daily for 2 weeks, followed by placebo or 300 mg bupropion once daily for subsequent 8 weeks (until week 22; visit 6) Second tapering placebo or 150 mg bupropion once daily for 7 days
  Interventions: Drug: Bupropion; Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — Crossover design: Oral administration of 150 mg bupropion once daily for 2 weeks, followed by 300 mg bupropion once daily for subsequent 8 weeks, tapering: 150 mg bupropion once daily for 7 days
  Other Names: Wellbutrin, Budeprion, Prexaton, Elontril, Aplenzin
Drug: Placebo — Crossover design: Oral administration of placebo once daily for 2 weeks, followed by placebo once daily for subsequent 8 weeks, tapering: placebo once daily for 7 days
  Other Names: control

SUMMARY:
The influence of bupropion compared to placebo on the change of apathy as quantified by the apathy evaluation scale (AES-I, where I [informant] is a friend or family member familiar with the daily activities of the subject) in patients with HD after ten (10) weeks of treatment.

DETAILED DESCRIPTION:
The safety and tolerability of Bupropion in HD.

The influence of Bupropion compared to placebo on the:

* change of apathy as quantified by the AES-C (clinician) or the AES-S (self),
* change of motor symptoms (UHDRS) and quantitative grip force motor assessment,
* change of cognitive symptoms (UHDRS and MMSE),
* change of psychiatric symptoms (UHDRS, HADS),
* change of activities of daily living (UHDRS),
* change of the NPI caregivers' distress score (NPI-D),
* change of ventral striatal and ventromedial prefrontal activation in response to a reward paradigm as quantified by fMRI.

ELIGIBILITY:
Inclusion Criteria:

1. Verified HD mutation carriers aged 25 to 75 years (inclusive) at first dosing
2. Apathetic as diagnosed by SCIA-D criteria
3. Stable concomitant medication (no change of medication during last six weeks prior to inclusion)
4. Written informed consent by prospective study participant before conduct of any trial-related procedure. Participant must be able to make an informed decision of whether or not to participate in the study
5. Patient has a caregiver (family member or friend), who is living in a close relationship with the patient and is willing to give written informed consent (caregiver) before performance of any trial-related procedure

Exclusion criteria:

1. Pregnant or nursing women
2. Active suicidality based on the answer "yes" in questions 4 and 5 of the Columbia-Suicide Severity Rating Scale (baseline version)
3. Woman of childbearing potential, not using highly effective methods of contraception defined as methods with a Pearl Index < 1 such as oral, topical or injected contraception, IUD, contraceptive vaginal ring, or double barrier method such as diaphragm and condom with spermicide) or not surgically sterile (via hysterectomy, ovariectomy or bilateral tubal ligation) or not at least one year post-menopausal
4. Male not using an acceptable barrier method for contraception and donating sperm from screening up to three months following treatment
5. Presence or history of any medically not controllable disease (e.g. uncontrolled arterial hypertension or diabetes mellitus)
6. Presence or history of seizures or diagnosed epilepsy or history of severe head trauma (contusion) or CNS tumor
7. Clinical significant renal (calculated creatine clearance < 60 ml/min) or hepatic dysfunction
8. Clinical significant depression defined by the NPI depression score (score ≥4 points) at screening
9. Schizophreniform psychosis within the last 6 months prior to first dose
10. History of anorexia or bulimia
11. Severe cognitive disorders defined as a score < 18 in the Mini- Mental State Examination (MMSE) at screening
12. Marked chorea (UHDRS 4) of face, BOL, trunk or extremities
13. Treatment with neuroleptics other than tiapride, MAO-B inhibitors, amantadine, levodopa, D- or D,L-amphetamine or psychostimulants like methylphenidate, modafinil or atomoxetine within 1 month prior to first dose
14. Known hypersensitivity reaction associated with bupropion, gelatine, lactose or magnesium stearate
15. Clinically relevant abnormal findings in the ECG, the vitals, in the physical examination or laboratory values at screening that could interfere with the objectives of the study or the safety of the subject as judged by the investigator
16. Acute disease state (e.g. nausea, vomiting, fever, diarrhoea, infection) within 7 days of first dose
17. Definite or suspected personal history or family history of adverse reactions or hypersensitivity to the trial compounds (or to compounds with a similar structure)
18. Presence of illicit drug and/or alcohol abuse
19. Participation in another investigative drug trial within 2 months or donation of blood within 12 weeks prior to the first dose or during the trial
20. Subjects who are unlikely to be compliant and attend scheduled clinic visits as required
21. Placement in an institution due to governmental or judicial authorities

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (AES-I) | 10 weeks
  The influence of Bupropion compared to placebo on the change of apathy as quantified by the apathy evaluation scale (AES-I, where I [informant] is a friend or family member familiar with the daily activities of the subject) in patients with HD after ten weeks of treatment.

SECONDARY OUTCOMES:
AES-C (clinician) | 10 weeks
  The influence of Bupropion compared to placebo on the change of apathy as quantified by the apathy evaluation scale (AES-C, where C [clinician] is the trial investigator) in patients with HD after ten weeks of treatment.
AES-S (self) | 10 weeks
  The influence of Bupropion compared to placebo on the change of apathy as quantified by the apathy evaluation scale (AES-S, where S [self] is the patient) in patients with HD after ten weeks of treatment.
Motor symptoms (UHDRS) | 10 weeks
  The influence of Bupropion compared to placebo on the UHDRS motor score in patients with HD after ten weeks of treatment.
Quantitative grip force motor assessment | 10 weeks
  The influence of Bupropion compared to placebo on motor scores in patients with HD after ten weeks of treatment.
Cognitive Symptoms | 10 weeks
  The influence of Bupropion compared to placebo on MMSE in patients with HD after ten weeks of treatment.
Psychiatric symptoms | 10 weeks
  The influence of Bupropion compared to placebo on UHDRS behavioural assessment in patients with HD after ten weeks of treatment.
Activities of daily living | 10 weeks
  The influence of Bupropion compared to placebo on UHDRS Functional Assessment in patients with HD after ten weeks of treatment.
Caregiver's distress | 10 weeks
  The influence of Bupropion compared to placebo on the NPI caregiver's distress score.
ventral striatal and ventromedial prefrontal activation | 10 weeks
  Change of ventral striatal and ventromedial prefrontal activation in response to a reward paradigm as quantified by fMRI.
Adverse events | 10 weeks
  The safety and tolerability of Bupropion will be compared with placebo in patients with HD after ten weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Priller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Neurologische Klinik der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum Ulm, Klinik für Neurologie, Ulm